CLINICAL TRIAL: NCT05042362
Title: A Double-blind, Randomized, Placebo-controlled Multicenter Study to Investigate Efficacy and Safety of Elinzanetant for the Treatment of Vasomotor Symptoms Over 26 Weeks in Postmenopausal Women
Brief Title: A Study to Learn More About How Well Elinzanetant Works and How Safe it is for the Treatment of Vasomotor Symptoms (Hot Flashes) That Are Caused by Hormonal Changes Over 26 Weeks in Women Who Have Been Through the Menopause
Acronym: OASIS-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21651; 2020-004908-33 (EudraCT Number)
Record Dates: First submitted 2021-08-26; First posted 2021-09-13 (Actual); Results first posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Vasomotor Symptoms Associated With Menopause; Hot Flashes
Keywords: Menopause
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Elinzanetant (BAY3427080) (Experimental): Participants will receive 120 mg elinzanetant orally once daily for 26 weeks.
  Interventions: Drug: Elinzanetant (BAY3427080)
- Placebo + elinzanetant (Placebo Comparator): Participants will receive matching placebo orally once daily for 12 weeks, followed by elinzanetant 120 mg for 14 weeks.
  Interventions: Drug: Elinzanetant (BAY3427080); Drug: Placebo

INTERVENTIONS:
Drug: Elinzanetant (BAY3427080) — 120 mg elinzanetant orally once daily
Drug: Placebo — Matching placebo orally once daily
  Arms: Placebo + elinzanetant

SUMMARY:
Researchers are looking for a better way to treat women who have hot flashes after women have been through the menopause. Hot flashes are caused by the hormonal changes that happen when a woman's body has been through the menopause. Menopause is when women stop having a menstrual cycle, also called a period. During the menopause, the ovaries increasingly produce less sex hormones as a result of the natural ageing process and related hormonal adjustments. The decline in hormone production can lead to various symptoms which, in some cases, can have a very adverse effect on a menopausal woman's quality of life.

The study treatment, elinzanetant, was developed to treat symptoms caused by hormonal changes. It works by blocking a protein called neurokinin from sending signals to other parts of the body, which is thought to play a role in starting hot flashes. There are treatments for hot flashes in women who have been through the menopause, but may cause medical problems for some people.

In this study, the researchers will learn how well elinzanetant works compared to a placebo in women who have been through the menopause and have hot flashes. A placebo looks like a treatment but does not have any medicine in it. To compare these study treatments, the doctors will ask the participants to record information about the participants' hot flashes in an electronic diary. The researchers will study the number of hot flashes the participants have and how severe the hot flashes are. The researchers will look at the results from before treatment, after 4 weeks, and after 12 weeks of treatment.

The participants in this study will take two capsules of either elinzanetant or the placebo once a day. The participants who take elinzanetant will take it for 26 weeks. The participants who take the placebo will take it for 12 weeks and then take elinzanetant for the next 14 weeks.

During the study, the participants will visit the site approximately 9 times and perform 1 visit by phone. Each participant will be in the study for approximately 36 weeks. The treatment duration will be 26 weeks.

During the study, the participants will:

* record information about the participants' hot flashes in an electronic diary
* answer questions about the participants' symptoms

The doctors will:

* check the participants' health
* take blood samples
* ask the participants questions about what medicines the participants are taking and if the participants are having adverse events An adverse event is any medical problem that a participant has during a study. Doctors keep track of all adverse events that happen in studies, even if doctors do not think the adverse events might be related to the study treatments.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal, defined as:

  1. at least 12 months of spontaneous amenorrhea prior to signing of informed consent, or
  2. at least 6 months of spontaneous amenorrhea prior to signing of informed consent with serum follicle-stimulating hormone (FSH) levels > 40 mIU/mL and a serum estradiol concentration of < 30 pg/mL, or
  3. at least 6 months after hysterectomy at signing of informed consent with serum FSH levels > 40 mIU/mL and a serum estradiol concentration of < 30 pg/mL, or
  4. surgical bilateral oophorectomy with or without hysterectomy at least 6 weeks prior to signing of informed consent.
* Moderate to severe hot flash (HF) associated with the menopause and seeking treatment for this condition.
* Participant has completed Hot Flash Daily Diary (HFDD) for at least 11 days during the two weeks preceding baseline visit, and participant has recorded at least 50 moderate or severe HF (including night-time HF) over the last 7 days that the HFDD was completed (assessed at the Baseline Visit).

Exclusion Criteria:

* Any clinically significant prior or ongoing history of arrhythmias, heart block and QT prolongation either determined through clinical history or on ECG evaluation.
* Any active ongoing condition that could cause difficulty in interpreting vasomotor symptoms (VMS) such as: infection that could cause pyrexia, pheochromocytoma, carcinoid syndrome.
* Current or history (except complete remission for 5 years or more) of any malignancy (except basal and squamous cell skin tumors). Women receiving adjuvant endocrine therapy (e.g. tamoxifen, aromatase inhibitors, GnRH analogues) cannot be enrolled in this study.
* Uncontrolled or treatment-resistant hypertension. Women with mild hypertension can be included in the study if these women are medically cleared prior to study participation.
* Untreated hyperthyroidism or hypothyroidism.

  * Treated hyperthyroidism with no abnormal increase of thyroid function laboratory parameters and no relevant clinical signs for > 6 months before signing of informed consent is acceptable.
  * Treated hypothyroidism with normal thyroid function test results during screening and a stable (for ≥ 3 months before signing of informed consent) dose of replacement therapy is acceptable.
* Any unexplained post-menopausal uterine bleeding.
* Clinically relevant abnormal findings on mammogram.
* Abnormal liver parameters.
* Disordered proliferative endometrium, endometrial hyperplasia, polyp, or endometrial cancer diagnosed based on endometrial biopsy during screening.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-11-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (99):
- United States (55):
  - Alabama Clinical Therapeutics | Birmingham, AL, Birmingham, Alabama
  - Central Research Associates | Birmingham, AL, Birmingham, Alabama
  - Mesa Obstetricians and Gynecologists | Research Department, Mesa, Arizona
  - MomDoc Women's Health Research | Scottsdale, AZ, Scottsdale, Arizona
  - Noble Clinical Research | Tucson, AZ, Tucson, Arizona
  - Del Sol Research | Women Health studies, Tucson, Arizona
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - Alliance Research Institute | Bell Gardens, CA, Bell Gardens, California
  - Diagnamics | Encinitas, CA, Encinitas, California
  - Om Research LLC | Lancaster, CA, Lancaster, California
  - Northern California Research | Sacramento, Sacramento, California
  - IntimMedicine | Washington, DC, Washington D.C., District of Columbia
  - AMR - Fort Myers, FL, Fort Myers, Florida
  - Suncoast Clinical Research Inc | Pinellas, Palm Harbor, Florida
  - Physician Care Clinical Research LLC | Sarasota, FL, Sarasota, Florida
  - Medisense Inc. | Atlanta, GA, Atlanta, Georgia
  - Paramount Research Solutions | College Park Location, College Park, Georgia
  - Soapstone Center for Clinical Research, Inc. | Decatur, GA, Decatur, Georgia
  - Drug Studies America, Marietta, Georgia
  - M3 Wake Research Atlanta, Sandy Springs, Georgia
  - Clinical Research Prime, Idaho Falls, Idaho
  - Investigators Research Group, LLC, Brownsburg, Indiana
  - The Iowa Clinic - Ankeny, Ankeny, Iowa
  - Southern Clinical Research Associates | Metairie, LA, Metairie, Louisiana
  - Continental Clinical Solutions | Towson, MD, Towson, Maryland
  - Revive Research Institute, Inc. - Women's Health, Dearborn Heights, Michigan
  - Valley OBGYN, Saginaw, Michigan
  - Women's Clinic of Lincoln, P.C. | Lincoln, NE, Lincoln, Nebraska
  - Jubilee Clinical Research Inc | Las Vegas, NV, Las Vegas, Nevada
  - Affiliated Clinical Research, Inc. | Las Vegas, NV, Las Vegas, Nevada
  - M3 Wake Research - Clinical Research Center of Nevada, Las Vegas, Nevada
  - The Center for Womens Health & Wellness, LLC | Lawrenceville, NJ, Lawrenceville, New Jersey
  - Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Velocity Clinical Research - Albuquerque, Albuquerque, New Mexico
  - Bosque Women's Care | Albuquerque, NM, Albuquerque, New Mexico
  - Circuit Clinical | OB GYN Associates of WNY, West Seneca, New York
  - OnSite Clinical Solutions - Charlotte, Charlotte, North Carolina
  - M3 Wake Research | Raleigh, NC, Raleigh, North Carolina
  - Unified Women's Clinical Research | Lyndhurst Clinical Research, Winston-Salem, NC, Winston-Salem, North Carolina
  - Axia Women's Health - Anderson Township, Cincinnati, Ohio
  - Centricity Research - Women's Health - Dublin, OH, Dublin, Ohio
  - HWC Women's Research Center | Englewood, OH, Englewood, Ohio
  - Hilltop Obstetrics & Gynecolofy, Franklin, Ohio
  - Women's Care Research Institute/Marion OBGYN, Inc., Marion, Ohio
  - University Hospitals | UH Cleveland Medical Center - MacDonald Clinical Trials Unit, Mayfield Heights, Ohio
  - Clinical Research Philadelphia | Philadelphia, PA, Philadelphia, Pennsylvania
  - MUSC Women's Health - Cannon St., Charleston, South Carolina
  - Venus Gynecology, LLC | Myrtle Beach, SC, Myrtle Beach, South Carolina
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Chattanooga Medical Research, LLC. | Chattanooga, TN, Chattanooga, Tennessee
  - Elligo Health Research | Women Partners in Health PLLC, Austin, Texas
  - Cedar Health Research, LLC. | DFW-East Clinical Site, Dallas, Texas
  - Maximos Ob/Gyn, League City, Texas
  - Northeast Clinical Research of San Antonio, LLC, San Antonio, Texas
  - Seattle Women's | Seattle, WA, Seattle, Washington
- Austria (5):
  - Medical University of Graz | Division of Gynecology and Obstetrics, Graz, Styria
  - Medizinische Universitat Innsbruck | Klinik fur Gyn Endokrinologie und Reproduktionsmedizin, Innsbruck, Tyrol
  - Kepler Campus IV | Gyn, Gburtshilfe & gyn. Endokrinologie, Linz, Upper Austria
  - AKH Wien | Allg. Gynaekologie & gynaekologische Onkologie, Vienna
  - Medizinische Universitat Wien | Universitatsklinik fur Frauenheilkunde Klinische Abteilung fur Gynakologische Endokrinologie, Vienna
- Czechia (10):
  - Gynekologie MEDA s.r.o., Brno
  - G-Centrum Olomouc s.r.o. Dr. Skrivanek, České Budějovice
  - GYN-MIKA s.r.o., České Budějovice
  - Gynekologie Cheb s.r.o., České Budějovice
  - MUDr. Stepan s.r.o., České Budějovice
  - GYN-F s.r.o., Hradec Králové
  - Kestr-gyn s.r.o., Náchod
  - PT-MEDICA s.r.o., Prachatice
  - GYNERA, Prague
  - Gynekologie Studentsky dum s.r.o., Prague
- Greece (7):
  - ARETAIEION University Hospital, Athens
  - University General Hospital of Athens "ATTIKON", Chaïdári
  - University General Hospital of Heraklion - Department of Paediatrics, Heraklion
  - Univ. General Hospital of Ioannina - Department of Paediatrics, Nephrology Unit, Ioannina
  - University General Hospital of Patras | Univ Obs & Gynae Cli, Pátrai
  - Hippokration General Hospital of Thessaloniki, Thessaloniki
  - General Hospital of Thessaloniki Papageorgiou, Thessaloniki
- Hungary (6):
  - TritonLife Medical Center, XIII.kerulet, Budapest
  - NAP-MED Egeszsegugyi Szolgaltato Kft, Debrecen
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Komaromi Selye Janos Korhaz, Komárom
  - SZTE ÁOK Szent Györgyi Albert Klinikai Kozpont, Szeged
  - Rub-Int Noi Egeszsegcentrum, Székesfehérvár
- Israel (6):
  - HaEmek Medical Center | Internal Medicine C Department - Research Unit, Afula
  - Mayanei HaYeshua Medical Center, Bnei Brak
  - Hillel Yaffe Medical Center, Hadera
  - Hadassah Hebrew University Hospital Ein Kerem, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Health Corporation of Galilee Medical Center, Nahariya
- Italy (7):
  - University Hospital Of Ferrara - Ostetricia e Ginecologia, Ferrara, Emilia-Romagna
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - Ospedale San Raffaele s.r.l. - Ginecologia Ostetricia e Medicina della Riproduzione, Milan, Lombardy
  - IRCCS Fondazione Policlinico San Matteo, Pavia, Lombardy
  - Azienda Ospedaliero-Universitaria Policlinico G. Rodolico-San Marco Di Catania, Catania, Sicily
  - Careggi University Hospital, Florence, Tuscany
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Tuscany
- Netherlands (3):
  - Flevoziekenhuis, Almere Stad
  - St. Antonius Ziekenhuis | Utrecht - R&D Interne Geneeskunde, Nieuwegein
  - Diakonessenhuis, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pinkerton JV, Simon JA, Joffe H, Maki PM, Nappi RE, Panay N, Soares CN, Thurston RC, Caetano C, Haberland C, Haseli Mashhadi N, Krahn U, Mellinger U, Parke S, Seitz C, Zuurman L. Elinzanetant for the Treatment of Vasomotor Symptoms Associated With Menopause: OASIS 1 and 2 Randomized Clinical Trials. JAMA. 2024 Aug 22;332(16):1343-54. doi: 10.1001/jama.2024.14618. Online ahead of print. PMID 39172446
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards. — https://clinicaltrials.bayer.com/study/21651
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217261&parentIdentifier=21651&attachmentIdentifier=2968ffc8-d6e1-4619-a54b-b0d8eea4f3d4&fileName=21651_PLS_English.pdf&versionIdentifier=
- See also: Study_Synopsis-21651.docx attachment has been generated from the Study Synopsis template. Data may be populated from the following (as available) : Study (44.0), Protocol (0.4), Results(0.1) — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217261&parentIdentifier=21651&attachmentIdentifier=d2ca5695-688e-4d2a-a610-90f3664b17b3&fileName=21651_Study_Synopsis_CTP.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 89 study centers in 8 countries, between 27-Aug-2021 (first participant first visit) and 27-Nov-2023 (last participant last visit).
Pre-assignment Details: A total of 1535 participants were screened; 1139 participants were not randomized. Most common reason for not being randomized was not meeting the eligibility criteria (1087 participants). 396 participants were randomized to treatment. A total of 197 participants were randomized to placebo - elinzanetant 120 mg arm and 199 participants to elinzanetant 120 mg arm.
Groups:
- Elinzanetant 120 mg: Participants received elinzanetant 120 mg orally once daily for 26 weeks.
- Placebo - Elinzanetant 120 mg: Participants received placebo for 12 weeks, followed by elinzanetant 120 mg orally once daily for 14 weeks.
Period: Overall Study
Arm/Group | Elinzanetant 120 mg | Placebo - Elinzanetant 120 mg
Started | 199 | 197
Completed | 154 | 155
Not Completed | 45 | 42
Not completed — Adverse Event | 7 | 9
Not completed — Lack of Efficacy | 0 | 2
Not completed — Lost to Follow-up | 7 | 4
Not completed — Missing | 4 | 2
Not completed — Withdrawal by Subject | 5 | 9
Not completed — Randomized by Mistake | 1 | 2
Not completed — Physician Decision | 3 | 0
Not completed — Other | 0 | 1
Not completed — Non-Compliance with Study Drug | 2 | 3
Not completed — incompleted treatment; finished follow-up | 16 | 10

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) was analyzed. FAS: all randomized subjects were included. Subjects in the full analysis set were analyzed according to the randomized intervention (intention-to-treat).
Groups:
- Total: Total of all reporting groups
Arm/Group | Elinzanetant 120 mg | Placebo - Elinzanetant 120 mg | Total
Number analyzed (Participants) | 199 | 197 | 396
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (4.9) | 54.5 (4.9) | 54.6 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 199 | 197 | 396
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 14 | 31
  Not Hispanic or Latino | 180 | 179 | 359
  Unknown or Not Reported | 2 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 38 | 38 | 76
  White | 151 | 154 | 305
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Frequency of Moderate to Severe HF From Baseline to Week 4 (Assessed by Hot Flash Daily Diary [HFDD]).
Description: The frequency of moderate to severe HF for each week during the treatment period was calculated using the available data during that particular week. Specifically for Week 4, Days 22-28 were used (Day 1 corresponds to start of treatment). Mean daily frequency is calculated as total number of moderate to severe HF during that week divided by the total number of available days with data during that week
Time Frame: From baseline to Week 4
Population: Participants in full analysis set (FAS) with evaluable data.
Measure: Mean (Standard Deviation); unit: Hot Flashes per day
Arm/Group | Elinzanetant 120 mg | Placebo - Elinzanetant 120 mg
Number analyzed (Participants) | 199 | 197
Hot Flashes per day
  Baseline | 13.38 (6.57) | 14.26 (13.94)
  Week 4: Change from baseline: number analyzed (Participants) | 191 | 185
  Week 4: Change from baseline | -7.48 (5.80) | -4.37 (6.73)
Statistical Analysis 1: Comparison: Elinzanetant 120 mg vs Placebo - Elinzanetant 120 mg; Test type: Superiority; p < 0.0001, Mixed model repeated measures (MMRM) — One-sided. A multiplicity adjustment strategy was defined using the graphical approach, controlling the overall type I error rate at a one-sided alpha level of 0.025 for confirmatory statistical superiority testing; Difference in LS-means = -3.29, 95% CI 2-sided [-4.47 to -2.10]

2. Primary Outcome: Mean Change in Frequency of Moderate to Severe HF From Baseline to Week 12 (Assessed by HFDD).
Description: The frequency of moderate to severe HF for each week during the treatment period was calculated using the available data during that particular week. Specifically for Week 12, Days 78-84 were used (Day 1 corresponds to start of treatment). Mean daily frequency is calculated as total number of moderate to severe HF during that week divided by the total number of available days with data during that week
Time Frame: From baseline to Week 12
Population: Participants in full analysis set (FAS) with evaluable data.
Measure: Mean (Standard Deviation); unit: Hot Flashes per day
Arm/Group | Elinzanetant 120 mg | Placebo - Elinzanetant 120 mg
Number analyzed (Participants) | 199 | 197
Hot Flashes per day
  Baseline | 13.38 (6.57) | 14.26 (13.94)
  Week 12: Change from baseline: number analyzed (Participants) | 175 | 169
  Week 12: Change from baseline | -8.74 (6.70) | -5.53 (10.16)
Statistical Analysis 1: Comparison: Elinzanetant 120 mg vs Placebo - Elinzanetant 120 mg; Test type: Superiority; p < 0.0001, MMRM — one-sided; Difference in LS-means = -3.22, 95% CI 2-sided [-4.81 to -1.63]

3. Primary Outcome: Mean Change in Severity of Moderate to Severe HF From Baseline to Week 4 (Assessed by HFDD).
Description: In the HFDD, hot flash (HF) severity is scored as 1=mild, 2=moderate, and 3=severe; a decrease indicates improvement. The diary records the number of mild, moderate, and severe HFs during day and night. Mild HFs are a "sensation of heat without sweating"; moderate are "heat with sweating but able to continue activity"; severe are "heat with sweating that stops activity."
  Baseline mean daily severity is calculated as:
  (2×moderateHFs+3×severeHFs)÷(totalmoderate+severeHFs).(2 × moderate HFs + 3 × severe HFs) ÷ (total moderate + severe HFs).(2×moderateHFs+3×severeHFs)÷(totalmoderate+severeHFs).
  If none occur, severity=0. Weekly severity during treatment is based on available days (Week 4: Days 22-28; Week 12: Days 78-84; Day 1=start of treatment), averaging the mean daily severity for that week. If more than 2 days are missing, the weekly value is set to missing.
Time Frame: From baseline to Week 4
Population: Participants in full analysis set (FAS) with evaluable data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Elinzanetant 120 mg | Placebo - Elinzanetant 120 mg
Number analyzed (Participants) | 199 | 197
Units on a scale
  Baseline | 2.56 (0.22) | 2.53 (0.23)
  Week 4: Change from baseline: number analyzed (Participants) | 191 | 185
  Week 4: Change from baseline | -0.73 (0.64) | -0.39 (0.43)
Statistical Analysis 1: Comparison: Elinzanetant 120 mg vs Placebo - Elinzanetant 120 mg; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 1, analysis 1]; Difference in LS-means = -0.33, 95% CI 2-sided [-0.44 to -0.23]

4. Primary Outcome: Mean Change in Severity of Moderate to Severe HF From Baseline to Week 12 (Assessed by HFDD).
Description: In the HFDD, hot flash (HF) severity is categorized as 1=mild, 2=moderate, 3=severe; thus, a decrease indicates improvement. The HFDD records the number of mild, moderate, and severe HFs during day and night. Mild HFs are a "sensation of heat without sweating"; moderate involve "heat with sweating but able to continue activity"; severe involve "heat with sweating that stops activity."
  Mean daily severity at baseline is calculated as:
  (2 × moderate HFs) + (3 × severe HFs)] ÷ (total moderate + severe HFs). If none occur, severity is set to 0. Weekly severity during treatment is based on available days (Week 4: Days 22-28; Week 12: Days 78-84; Day 1=start of treatment), averaging mean daily severity across that week. If more than 2 days are missing, the week is set to missing.
Time Frame: From baseline to Week 12
Population: Participants in full analysis set (FAS) with evaluable data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Elinzanetant 120 mg | Placebo - Elinzanetant 120 mg
Number analyzed (Participants) | 199 | 197
Units on a scale
  Baseline | 2.56 (0.22) | 2.53 (0.23)
  Week 12: Change from baseline: number analyzed (Participants) | 175 | 169
  Week 12: Change from baseline | -0.95 (0.78) | -0.55 (0.60)
Statistical Analysis 1: Comparison: Elinzanetant 120 mg vs Placebo - Elinzanetant 120 mg; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 1, analysis 1]; Difference in LS-means = -0.40, 95% CI 2-sided [-0.54 to -0.25]

5. Secondary Outcome: Mean Change in Frequency of Moderate to Severe HF From Baseline to Week 1 (Assessed by HFDD).
Description: The frequency of moderate to severe HF for each week during the treatment period was calculated using the available data during that particular week. Specifically for Week 1, Days 2-8 were used (Day 1 corresponds to start of treatment). Mean daily frequency is calculated as total number of moderate to severe HF during that week divided by the total number of available days with data during that week
Time Frame: From baseline to Week 1
Population: Participants in full analysis set (FAS) with evaluable data.
Measure: Mean (Standard Deviation); unit: Hot Flashes per day
Arm/Group | Elinzanetant 120 mg | Placebo - Elinzanetant 120 mg
Number analyzed (Participants) | 199 | 197
Hot Flashes per day
  Baseline | 13.38 (6.57) | 14.26 (13.94)
  Week 1: Change from baseline: number analyzed (Participants) | 196 | 189
  Week 1: Change from baseline | -5.00 (5.05) | -2.72 (4.99)
Statistical Analysis 1: Comparison: Elinzanetant 120 mg vs Placebo - Elinzanetant 120 mg; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 1, analysis 1]; Difference in LS-means = -2.45, 95% CI 2-sided [-3.36 to -1.55]

6. Secondary Outcome: Mean Change in Frequency of Moderate to Severe HF From Baseline Over Time.
Description: The frequency of moderate to severe HF for each week during the treatment period was calculated using the available data during that particular week. Specifically, for Week 1 Days 2-8 were used instead of 1-7, because the intake started on Day 1 only before going to bed, for Week 4 Days 22-28 were used and for Week 12 Days 78-84 were used (Day 1 corresponds to start of treatment). These data were aggregated to a mean daily frequency as (total number of moderate to severe HF during that week) / (total number of available days with data during that week). In case data was not available for more than 2 days within a week, the value for that particular week was set to missing.
Time Frame: From baseline to Week 30
Population: Participants in full analysis set (FAS) with evaluable data.
Measure: Mean (Standard Deviation); unit: Hot Flashes per day
Arm/Group | Elinzanetant 120 mg | Placebo - Elinzanetant 120 mg
Number analyzed (Participants) | 199 | 197
Hot Flashes per day
  Baseline | 13.38 (6.57) | 14.26 (13.94)
  Week 1: Change from baseline: number analyzed (Participants) | 196 | 189
  Week 1: Change from baseline | -5.00 (5.05) | -2.72 (4.99)
  Week 4: Change from baseline: number analyzed (Participants) | 191 | 185
  Week 4: Change from baseline | -7.48 (5.8) | -4.37 (6.73)
  Week 8: Change from baseline: number analyzed (Participants) | 180 | 175
  Week 8: Change from baseline | -8.42 (6.5) | -5.24 (8.08)
  Week 12: Change from baseline: number analyzed (Participants) | 175 | 169
  Week 12: Change from baseline | -8.74 (6.7) | -5.53 (10.16)
  Week 16: Change from baseline: number analyzed (Participants) | 170 | 160
  Week 16: Change from baseline | -9.19 (6.21) | -8.08 (8.87)
  Week 20: Change from baseline: number analyzed (Participants) | 161 | 160
  Week 20: Change from baseline | -9.87 (6.40) | -8.88 (8.30)
  Week 26: Change from baseline: number analyzed (Participants) | 114 | 110
  Week 26: Change from baseline | -10.11 (6.41) | -10.10 (8.75)
  Week 30: Change from baseline: number analyzed (Participants) | 141 | 129
  Week 30: Change from baseline | -6.70 (5.99) | -6.15 (10.52)

7. Secondary Outcome: Mean Change in Patient-reported Outcomes Measurement Information System Sleep Disturbance Short Form 8b (PROMIS SD SF 8b) Total T-score From Baseline to Week 12.
Description: In controversy of what you have been proposing above here you are just explaining the PROMIS SD SF 8b scores, not the secondary endpoint which is the change in the T-scores from BL to week 12
  The PROMIS Sleep Disturbance Short Form 8b (PROMIS SD SF 8b) measures sleep disturbance over the past 7 days using 8 items assessing sleep quality, depth, restorative sleep, difficulty falling or staying asleep, and perceptions of sleep adequacy and satisfaction. Items use 5-point response options that vary by item (e.g., Not at all → Very much; Never → Always; Very poor → Very good). Item scores sum to a raw score of 8-40, which is converted to a T-score (mean 50, SD 10; range 28.9-76.5). Higher scores reflect greater sleep disturbance. PROMIS cut points classify T-scores of 55-59 as mild, 60-69 as moderate, and ≥70 as severe disturbance.
Time Frame: From baseline to Week 12
Population: Participants in full analysis set (FAS) with evaluable data.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Elinzanetant 120 mg | Placebo - Elinzanetant 120 mg
Number analyzed (Participants) | 199 | 197
T-score
  Baseline: number analyzed (Participants) | 184 | 179
  Baseline | 61.0 (7.7) | 60.2 (7.2)
  Week 12: Change from baseline: number analyzed (Participants) | 166 | 156
  Week 12: Change from baseline | -10.8 (9.6) | -5.0 (6.9)
Statistical Analysis 1: Comparison: Elinzanetant 120 mg vs Placebo - Elinzanetant 120 mg; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 1, analysis 1]; Difference in LS-means = -5.58, 95% CI 2-sided [-7.18 to -3.98]

8. Secondary Outcome: Mean Menopause Specific Quality of Life Scale (MENQOL) Total Score From Baseline to Week 12.
Description: The MENQOL questionnaire was comprised of 29 items assessing the presence of menopausal symptoms and the impact of menopause on health-related quality of life over the past week. The items assessed four domains of symptoms and functioning: VMS, psychosocial functioning, physical functioning, and sexual functioning. For each item, the participant indicated if they had experienced the symptom (yes/no). If participants selected yes, participants rated how bothered they were by the symptom using a six-point verbal descriptor scale, with response options ranging from 0 'not at all bothered' to 6 'extremely bothered'. Based on the individual responses, item scores, domain scores, and a total MENQOL score were calculated. Each score ranged from 1-8, higher scores indicated greater bother.
Time Frame: From baseline to Week 12
Population: Participants in full analysis set (FAS) with evaluable data.
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Elinzanetant 120 mg | Placebo - Elinzanetant 120 mg
Number analyzed (Participants) | 199 | 197
Scores on scale
  Baseline: number analyzed (Participants) | 179 | 173
  Baseline | 4.56 (1.27) | 4.49 (1.31)
  Week 12: Change from baseline: number analyzed (Participants) | 160 | 152
  Week 12: Change from baseline | -1.41 (1.30) | -0.96 (1.11)
Statistical Analysis 1: Comparison: Elinzanetant 120 mg vs Placebo - Elinzanetant 120 mg; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 1, analysis 1]; Difference in LS-means = -0.42, 95% CI 2-sided [-0.64 to -0.20]

9. Secondary Outcome: Mean Beck Depression Inventory (BDI-II) Total Score From Baseline to Week 12.
Description: The BDI-II was a 21-item questionnaire assessed the intensity of depressive symptoms over the past 2 weeks. Each item was a list of four statements arranged in increasing levels of severity about a particular symptom of depression. Items used a 4-point verbal response scale ranging from 0 (not at all) to 3 (extreme form of each symptom); specific response options were tailored to the aspect of depression being measured in each item. A total score ranging from 0 to 63 was calculated with scores of 0-13 indicating mild minimal range, 14 - 19 mild depression, 20 - 28 indicating moderate and 29 - 63 severe depression (higher score = greater depression).
Time Frame: From baseline to Week 12
Population: Participants in full analysis set (FAS) with evaluable data.
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Elinzanetant 120 mg | Placebo - Elinzanetant 120 mg
Number analyzed (Participants) | 199 | 197
Scores on scale
  Baseline | 6.8 (6.5) | 6.2 (6.7)
  Week 12: Change from baseline: number analyzed (Participants) | 175 | 168
  Week 12: Change from baseline | -0.5 (7.2) | 0.9 (6.5)

10. Secondary Outcome: Mean Change in BDI-II Total Score From Baseline to Week 26.
Description: The BDI-II was a 21-item questionnaire assessing the intensity of depressive symptoms over the past 2 weeks. Each item was a list of four statements arranged in increasing levels of severity about a particular symptom of depression. Items used a 4-point verbal response scale ranging from 0 (not at all) to 3 (extreme form of each symptom); specific response options were tailored to the aspect of depression being measured in each item. A total score ranging from 0 to 63 was calculated with scores of 0-13 indicating mild minimal range, 14 - 19 mild depression, 20 - 28 indicating moderate and 29 - 63 severe depression (higher score = greater depression).
Time Frame: From baseline to Week 26
Population: Participants in full analysis set (FAS) with evaluable data.
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Elinzanetant 120 mg | Placebo - Elinzanetant 120 mg
Number analyzed (Participants) | 199 | 197
Scores on scale
  Baseline | 6.8 (6.5) | 6.2 (6.7)
  Week 26: Change from baseline: number analyzed (Participants) | 108 | 104
  Week 26: Change from baseline | -0.9 (6.7) | -0.6 (5.5)

ADVERSE EVENTS:
Time Frame: From the start of study medication up to 14 days after the last dose of medication, approximately 28 weeks. Adverse event reporting for the all-cause mortality considers all deaths that occurred at any time during the study before the last contact, approximately 30 weeks.
Groups:
- Elinzanetant 120 mg Week 1-12: Subjects who received elinzanetant 120 mg during Weeks 1-12. Reported AEs for the exposure period Weeks 1-12 to elinzanetant.
- Placebo Week 1-12: Subjects who received placebo during Weeks 1-12. Reported AEs for the exposure period to placebo.
- Elinzanetant 120 mg Week 13-26: Subjects who received elinzanetant 120 mg during Weeks 1-12 and continued with elinzanetant 120 mg after Week 12. Reported AEs for the exposure period Weeks 13 - 26 to elinzanetant.
- Placebo - Elinzanetant 120 mg Week 13-26: Subjects who received placebo during Weeks 1-12 and switched to elinzanetant 120 mg after Week 12. Reported AEs for the exposure period to elinzanetant.
- Elinzanetant 120 mg Week 1-26: Subjects who received elinzanetant 120 mg at any time during the study (including those who switched from placebo to elinzanetant 120 mg at Week 13). Reported AEs for the exposure period to elinzanetant for both treatment groups.
Arm/Group | Elinzanetant 120 mg Week 1-12 | Placebo Week 1-12 | Elinzanetant 120 mg Week 13-26 | Placebo - Elinzanetant 120 mg Week 13-26 | Elinzanetant 120 mg Week 1-26
All-Cause Mortality (participants affected / at risk) | 0/199 | 0/194 | 0/171 | 0/168 | 0/367
Serious Adverse Events (participants affected / at risk) | 4/199 | 2/194 | 0/171 | 9/168 | 13/367
Other Adverse Events (participants affected / at risk) | 38/199 | 28/194 | 6/171 | 9/168 | 51/367
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elinzanetant 120 mg Week 1-12 (N=199) | Placebo Week 1-12 (N=194) | Elinzanetant 120 mg Week 13-26 (N=171) | Placebo - Elinzanetant 120 mg Week 13-26 (N=168) | Elinzanetant 120 mg Week 1-26 (N=367)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthrodesis (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bunion operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Mammoplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elinzanetant 120 mg Week 1-12 (N=199) | Placebo Week 1-12 (N=194) | Elinzanetant 120 mg Week 13-26 (N=171) | Placebo - Elinzanetant 120 mg Week 13-26 (N=168) | Elinzanetant 120 mg Week 1-26 (N=367)
Fatigue (General disorders) | 14 (14) | 3 (3) | 0 (0) | 1 (1) | 15 (15)
Depression rating scale score increased (Investigations) | 12 (13) | 11 (12) | 1 (1) | 2 (2) | 14 (16)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (10) | 10 (11) | 1 (1) | 1 (1) | 12 (12)
Headache (Nervous system disorders) | 14 (14) | 5 (5) | 4 (4) | 6 (7) | 24 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI will submit any proposed publications to the sponsor, who may advise PI within 30 days of any information that is confidential or requires protection and may request to remove confidential information or delay the publication for 60 days. For this multicenter study, PI will not, without the sponsor's consent, publish results until a multicenter publication is published; if that is not done within 12 months after study completion, PI may publish results in accordance with above provisions.

DOCUMENTS (2):
  • Study Protocol (2022-06-22): https://cdn.clinicaltrials.gov/large-docs/62/NCT05042362/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-07): https://cdn.clinicaltrials.gov/large-docs/62/NCT05042362/SAP_001.pdf